CLINICAL TRIAL: NCT02845219
Title: A Trial Investigating the Influence of Oral Semaglutide on Pharmacokinetics of Ethinylestradiol and Levonorgestrel in an Oral Contraceptive Combination Drug in Healthy Postmenopausal Females
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN9924-4249; 2015-004232-35 (EudraCT Number); U1111-1174-7914 (Other: WHO)
Record Dates: First submitted 2016-07-13; First posted 2016-07-27 (Estimated); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — semaglutide; ethinyl estradiol, levonorgestrel drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oral contraceptive/SNAC/Oral Trial drug (Experimental)
  Interventions: Drug: semaglutide; Drug: SNAC; Drug: Microgynon®

INTERVENTIONS:
Drug: semaglutide — Oral administration once daily alone or together with oral contraceptive.
Drug: SNAC — Oral administration once daily together with oral contraceptive.
Drug: Microgynon® — Oral administration once daily alone or together with oral semaglutide or SNAC.

SUMMARY:
This trial is conducted in Europe. The aim of the trial is to investigate the influence of oral semaglutide on pharmacokinetics (the exposure of the trial drug in the body) of ethinylestradiol and levonorgestrel in an oral contraceptive combination drug in healthy postmenopausal females.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal female, age at least 45 years at the time of signing informed consent. With at least 12 consecutive months since the last spontaneous menstrual bleeding (if there was any uncertainty of the time of the last spontaneous bleeding, the postmenopausal status is to be confirmed with follicle stimulating hormone (FSH) 40 mIU/mL)
* Body mass index (BMI) between 20.0 and 29.9 kg/m^2 (both inclusive)
* Considered to be generally healthy based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator

Exclusion Criteria:

* Smoker (defined as a subject who is smoking at least one cigarette or the equivalent per day). A subject smoking less than one cigarette or the equivalent per day must be able or willing to refrain from smoking and use of nicotine substitute products during the trial
* Any blood draw in excess of 25 mL in the past 30 days, or donation of blood or plasma in excess of 400 mL within the 90 days preceding screening
* Sitting blood pressure at screening (after resting for at least 5 minutes) outside the range of 90-139 mmHg for systolic or 50-89 mmHg for diastolic. If white-coat hypertension is suspected a single repeat measurement is allowed, last measurement being conclusive
* History of major surgical procedures involving the stomach potentially affecting absorption of trial product (e.g. subtotal and total gastrectomy, sleeve gastrectomy, gastric bypass surgery)

Min Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Area under the ethinylestradiol plasma concentration-time curve during a dosing interval (0-24 hours) at steady state | On day 8 (OC alone), day 24 (OC with SNAC) and day 82 (OC with oral semaglutide at steady state)
Area under the levonorgestrel plasma concentration-time curve during a dosing interval (0-24 hours) at steady state | On day 8 (OC alone), day 24 (OC with SNAC) and day 82 (OC with oral semaglutide at steady state)

SECONDARY OUTCOMES:
Maximum observed ethinylestradiol plasma concentration during a dosing interval (0-24 hours) at steady state | On day 8 (OC alone), day 24 (OC with SNAC) and day 82 (OC with oral semaglutide at steady state)
Maximum observed levonorgestrel plasma concentration during a dosing interval 0-24 hours) at steady state | On day 8 (OC alone), day 24 (OC with SNAC) and day 82 (OC with oral semaglutide at steady state)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Berlin, Germany

REFERENCES:
- [Derived] Jordy AB, Albayaty M, Breitschaft A, Anderson TW, Christiansen E, Houshmand-Oregaard A, Manigandan E, Baekdal TA. Effect of Oral Semaglutide on the Pharmacokinetics of Levonorgestrel and Ethinylestradiol in Healthy Postmenopausal Women and Furosemide and Rosuvastatin in Healthy Subjects. Clin Pharmacokinet. 2021 Sep;60(9):1171-1185. doi: 10.1007/s40262-020-00976-x. PMID 33782832
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com